CLINICAL TRIAL: NCT05464212
Title: Comparison of the Efficacy of Ultrasound-guided Greater Occipital Nerve Block and Pulsed Radiofrequency Therapy in Chronic Migraine Patients: A Randomized Controlled Double-Blind Study
Brief Title: Comparison of the Efficacy of Ultrasound-guided Greater Occipital Nerve Block and Pulsed Radiofrequency Therapy in Chronic Migraine Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Tuba Tanyel, Medical Doctor, Research Assistant, Eskisehir Osmangazi University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ESOGU-TTANYEL-01
Record Dates: First submitted 2022-07-05; First posted 2022-07-19 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Chronic Migraine, Headache
MeSH Terms: conditions — Headache

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- USG Guided Greater Occipital Nerve Block (GONB) (Active Comparator)
  Interventions: Procedure: USG Guided Greater Occipital Nerve Block
- USG Guided Greater Occipital Nerve Block and Pulsed Radiofrequency (GONB+PRF) (Active Comparator)
  Interventions: Procedure: USG Guided Greater Occipital Nerve Block and Pulsed Radiofrequency

INTERVENTIONS:
Procedure: USG Guided Greater Occipital Nerve Block — With 0.5 Hz sensorial stimulation, a 5-cm-long radiofrequency needle with a 0.5 cm active tip was advanced under ultrasound guidance in both pulsed PRF and nerve block groups. USG probe was located to medial one-third of the superior nuchal line between the occipital tubercle and mastoid process under sterile conditions. Finally, the placement of the needle was verified by Doppler imaging of the occipital artery. A 0.3-0.5 Hz sensory stimulus was given with the RF device, and the paresthesia sensation in the patient's occipital nerve dermatome was questioned, and location verification was performed. Then, GON block was performed in all patients by administering 5mg bupivacaine through a PRF needle. After the GON block, the PRF neuromodulation was applied at 42 degrees for 4 minutes in the GONB-PRF group. In the GONB group, the PRF generator was set for 4 minutes, and the time was waited, but no pulse was given.
  Arms: USG Guided Greater Occipital Nerve Block (GONB)
Procedure: USG Guided Greater Occipital Nerve Block and Pulsed Radiofrequency — With 0.5 Hz sensorial stimulation, a 5-cm-long radiofrequency needle with a 0.5 cm active tip was advanced under ultrasound guidance in both pulsed PRF and nerve block groups. USG probe was located to medial one-third of the superior nuchal line between the occipital tubercle and mastoid process under sterile conditions. Finally, the placement of the needle was verified by Doppler imaging of the occipital artery. A 0.3-0.5 Hz sensory stimulus was given with the RF device, and the paresthesia sensation in the patient's occipital nerve dermatome was questioned, and location verification was performed. Then, GON block was performed in all patients by administering 5mg bupivacaine through a PRF needle. After the GON block, the PRF neuromodulation was applied at 42 degrees for 4 minutes in the GONB-PRF group. In the GONB group, the PRF generator was set for 4 minutes, and the time was waited, but no pulse was given.
  Arms: USG Guided Greater Occipital Nerve Block and Pulsed Radiofrequency (GONB+PRF)

SUMMARY:
Chronic migraine (CM) is related to headache-related disability and reduced quality of life. Therefore, patients with CM require preventive treatment. The aim of this double-blind, comparative-effectiveness study was to compare ultrasound-guided great occipital nerve (GON) block and pulsed radiofrequency (PRF) application in CM patients.

The study consisted of 2 groups: GON block (group GONB) and GON block + pulsed RF (group GONB+PRF). Each group had 16 patients. Ultrasound-guided GONB was performed to locate the nerve more accurately. With 0.5 Hz sensorial stimulation, a 5-cm-long radiofrequency needle was advanced under ultrasound guidance in both groups. GON block was performed in all patients by administering 5mg bupivacaine through a PRF needle. After the GON block, the PRF neuromodulation was applied at 42 degrees for 4 minutes in the GONB-PRF group. In the GONB group, no pulse was given. The patients were examined for follow-ups at the 1st, 2nd, 3rd, and 6th months after the procedure. The severity and the number of migraine attacks, and the number of analgesic drugs were noted.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65;
* ICHD-3 defined chronic migraine

Exclusion Criteria:

* Patients who had been started on an effective preventive medication within the past three months;
* Medication-overuse headache;
* Treatment with peripheral nerve blocks, trigger point injections or botulinum toxin injections within the past three months;
* Known allergic reaction to local anaesthetics;
* Pregnancy or nursing;
* History of another headaches;
* History of chronic medical conditions (e.g. cardiovascular, hepatic, renal, endocrine);
* History of other chronic pain syndromes (e.g. low back pain and fibromyalgia).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2019-10-20 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Visuel Analog Scale | 6 months
  The lowest score on the visual analog scale is 0 and the highest score is 10. 10 indicates very severe pain, 0 indicates no pain

CONTACTS AND LOCATIONS:
Locations (1):
- Eskisehir Osmangazi University, Eskişehir, Odunpazari, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tanyel Saracoglu T, Bilir A, Gulec MS. Effectiveness of combining greater occipital nerve block and pulsed radiofrequency treatment in patients with chronic migraine: a double-blind, randomized controlled trial. Head Face Med. 2024 Sep 11;20(1):48. doi: 10.1186/s13005-024-00449-7. PMID 39256847

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-04-30): https://cdn.clinicaltrials.gov/large-docs/12/NCT05464212/Prot_SAP_000.pdf
  • Informed Consent Form (2019-04-30): https://cdn.clinicaltrials.gov/large-docs/12/NCT05464212/ICF_001.pdf